CLINICAL TRIAL: NCT03881800
Title: Population Pharmacokinetics and Dosing Regimens Optimization of Ceftazidime in Critically Ill Burn Children
Brief Title: Ceftazidime in Burn Children
Acronym: CEFTAZOPTIM
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP180163; 2019-A00035-52 (Other: ID-RCB)
Record Dates: First submitted 2019-02-18; First posted 2019-03-20 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Burned Children; Ceftazidime Treatment
Keywords: Ceftazidime; Burned Children; Intensive care; Pharmacokinetic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: titration- blood sample — Ceftazidime titration

SUMMARY:
Concentrations and effects of Ceftazidime in critically ill burn children are unpredictable and the risk of under-exposure may be associated with poor clinical outcomes. In addition, between-subject variability (BSV) is known to be substantial in critically ill burn children.

Optimization of Ceftazidime dosing is therefore desirable for all. The investigators aim to investigate, using a population approach, the pharmacokinetics (PK) of Ceftazidime including PK/pharmacodynamic (PD) targets (fT(%) > minimal inhibitory concentration (MIC)) and PD endpoints (clinical outcomes) in critically ill burn children. The effects of covariates on Ceftazidime PK and PK/PDs are investigated in order to better explain the BSV and to ultimately suggest individualized dosage regimens.

It will be a prospective PK study. Six blood samples were taken from each patient during dosing interval. The primary PK/ PD targets were Ceftazidime concentrations above the MIC of the pathogen at both 50% (50% f T>MIC) and 100% (100% f T>MIC) of the dosing interval. The investigators used skewed logistic regression to describe the effect of Ceftazidime exposure on patient outcome.

DETAILED DESCRIPTION:
Background and aims of the study:

Recent studies have suggested a risk of under-exposure to anti-infectives in critically ill adults. This under-exposure may be associated with poor clinical outcomes as well as a delay or incomplete clinical resolution of infection; The dosing regimen of anti-infectives in critically ill children is usually based on weight (i.e. mg per Kg). However, between-subject variability is known to be substantial in children and even more so with burns and in critical illness. Ceftazidime is one of the most anti-infective agents used in this vulnerable population. Given to the expected high BSV, concentrations and effects of Ceftazidime are unpredictable and the risk of under exposure- is thus considerable. Rationalization of Ceftazidime in children is therefore desirable.

The purpose of the present study is to investigate, using a population approach, the pharmacokinetics (PK) and pharmacodynamics (PD) of Ceftazidime including usual PK/PD targets (fT(%) > minimal inhibitory concentration (MIC)) and PD endpoints (clinical outcomes) in critically ill burn children. The effects of developmental and other factors related to critical illness and burns on Ceftazidime PK and PK/PDs are investigated in order to better explain the observed between-subject variabilities and to ultimately suggest individualized dosage regimens.

This prospective study will be conducted in a paediatric intensive care unit of Public Hospitals in Paris, France

Intervention:

Patient selection will take place in paediatric intensive care unit. The senior physician proposes the study to holders of parental authority whose child receives or will receive Ceftazidime during its follow-up or hospitalization.

The senior physician will give a briefing note to the holders of parental authority, and if the child is able to understand the information. The non-oral opposition for the retrieval and analysis of data will be collected.

No intervention or no charge will be made for this study

ELIGIBILITY:
Inclusion Criteria:

* Patient age: > 1 month and < 18 years
* Patient weight > 3 Kg
* Patient requiring the administration of Ceftazidime for the treatment of a documented or suspected bacterial infection

Exclusion Criteria:

* Patient and parents having notified to the doctor that they refuse data recovery and additional blood sample volume

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Burned children requiring the administration of Ceftazidime for the treatment of a documented or suspected bacterial infection
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2020-11-11 (Actual)

PRIMARY OUTCOMES:
Ceftazidime concentration | Up to 28 days
  6 blood samples

SECONDARY OUTCOMES:
Weight (kg) | Up to 28 days
  Composite measure of the health condition : clinical data
Body temperature (°C) | Up to 28 days
  Composite measure of the health condition : clinical data
Creatinine clearance | Up to 28 days
  Composite measure of the health condition : biological data
Albumin levels | Up to 28 days
  Composite measure of the health condition : biological data
PELOD-2 score (severity score) | Up to 28 days
  Composite measure of the health condition : clinical data
Percentage of body surface burned | Up to 28 days
  Composite measure of the health condition : clinical data
C Reactive Protein | Up to 28 days
  Composite measure of the health condition : biological data
Relapse | Day 28 after end of Ceftazidime administration
  Composite measure of the health condition
Minimum Inhibitory Concentration (MIC) of the suspected or documented pathogen | Day 28 after end of Ceftazidime administration

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi OUALHA, MD PhD, Principal Investigator — Hospital Necker - Enfants Malades
Locations (1):
- Hospital Necker - Enfants Malades (Public Hospitals of Paris), Paris, France

IPD SHARING:
Plan to Share IPD: No